CLINICAL TRIAL: NCT07262528
Title: Hand Rehabilitation in People With Hemiparesis After a Stroke Using 3D Imaging With fNIRS Neurofeedback
Brief Title: fNIRS Neurofeedback for Post-stroke Hand Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Agnieszka Guzik, PhD, Principal Investigator, University of Rzeszow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8/01/2020
Record Dates: First submitted 2025-09-28; First posted 2025-12-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Rehabilitation supplemented with Biofeedback HEG (Experimental)
  Interventions: Other: Standard Rehabilitation supplemented with Biofeedback HEG
- Control: Standard Rehabilitation (Other)
  Interventions: Other: Standard Rehabilitation

INTERVENTIONS:
Other: Standard Rehabilitation supplemented with Biofeedback HEG — The experimental group will be provided with rehabilitation at the Rehabilitation Clinic and additional exercises with Biofeedback HEG. HEG therapy will be conducted for 15 days, every day from Monday to Friday. The duration of one session is 30 minutes. The HEG Neurofeedback therapy equipment will be supplemented with new hand therapy software. During the exercises, patients will focus on a discussed and presented task, and once the expected level of concentration is reached, the software will trigger a virtual hand performing a finger flexion movement.
  Arms: Standard Rehabilitation supplemented with Biofeedback HEG
Other: Standard Rehabilitation — Participants from the control group will be provided with rehabilitation at the Rehabilitation Clinic and an additional 30 minutes of individual physiotherapy focused on restoring hand function.
  Arms: Control: Standard Rehabilitation

SUMMARY:
Cardiovascular diseases are one of the main causes of disability. Among post-stroke individuals, 80% experience upper limb dysfunction, while only 5% to 20% of individuals regain full limb and hand function. The purpose of this study is to evaluate the effects of hand rehabilitation of post-stroke individuals using HEG Neurofeedback The study will include 30 participants in the early sub-acute phase post-stroke, who will be assigned to either the study group or the control group. Participants in the experimental group will follow a rehabilitation program extended with HEG Neurofeedback training, while participants in the control group will follow the standard rehabilitation program.

The HEG Neurofeedback therapy equipment will be supplemented with new hand therapy software. During the exercises, patients will focus on a discussed and presented task, and once the expected level of concentration is reached, the software will trigger a virtual hand performing a finger flexion movement.

Motor control of the hand will be assessed using the Fugl-Meyer Scale and Brunnström recovery stages.

DETAILED DESCRIPTION:
This study is a prospective, randomized, single-blind clinical trial with intervention. Participants will be recruited from among patients treated at the Rehabilitation Clinic. Inclusion criteria: individuals with hemiparesis after a first ischemic stroke, subacute stroke period (no longer than 3 months), upper limb paresis rated 2-4 by Brunnstrom recovery stages, participants aged 18 to 70 years, consent to participate in the study. Exclusion criteria: unstable general condition, visual field disorders, inability to sit independently, cognitive impairment (Mini-Mental State Examination, MMSE > 24). The minimum size of the sample was calculated taking into account the number of individuals after stroke hospitalized annually in the re habilitation ward, i.e. approximately 120 patients, of which those in the acute phase of recovery constitute about 40%. It was assumed that 80% of the patients would have a minimum 2 in Brunnstrom scale. A fraction size of 0.8 was used, with a maximum error of 5%, a sample size of 30 patients was obtained.

The allocation of interventions will be determined based on a simple randomization sequence generated using Microsoft Excel. The study coordinator will register participants, generate the random allocation sequence, and assign and schedule participants for the interventions.

Fifteen participants will be assigned to the experimental group and fifteen to the control group.

Interwention. The experimental group will be provided with rehabilitation at the Rehabilitation Clinic and additional exercises with Biofeedback HEG. HEG therapy will be conducted for 15 days, every day from Monday to Friday. The duration of one session is 30 minutes. Participants from the control group will be provided with rehabilitation at the Rehabilitation Clinic and an additional 30 minutes of individual physiotherapy focused on restoring hand function.

Participants will be assessed twice, before the start of the therapy series and immediately after its completion. Motor control of the hand will be assessed using the Fugl-Meyer Scale and Brunnström recovery stages.

ELIGIBILITY:
Inclusion Criteria:

* individuals with hemiparesis after a first ischemic stroke,
* subacute stroke period (no longer than 3 months),
* upper limb paresis rated 2-4 by Brunnstrom recovery stages,
* participants aged 18 to 70 years,
* consent to participate in the study.

Exclusion Criteria:

* unstable general condition,
* visual field disorders,
* inability to sit independently,
* cognitive impairment (Mini-Mental State Examination, MMSE > 24).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Hand motor control - Fugl-Meyer Assessment (Upper Limb, Wrist, and Hand Section) | Baseline (Day 1)
  Assessment will be performed using the Fugl-Meyer Assessment for the upper limb, including wrist and hand function, to evaluate motor recovery after stroke. The wrist section has a minimum score of 0 and a maximum score of 10, while the hand section has a minimum score of 0 and a maximum score of 14. In both sections, higher scores indicate better motor function.
Hand motor control - Fugl-Meyer Assessment (Upper Limb, Wrist, and Hand Section) | Immediately after therapy completion (Day 15)
  Assessment will be performed using the Fugl-Meyer Assessment for the upper limb, including wrist and hand function, to evaluate motor recovery after stroke. The wrist section has a minimum score of 0 and a maximum score of 10, while the hand section has a minimum score of 0 and a maximum score of 14. In both sections, higher scores indicate better motor function.
Hand motor control - Brunnström Recovery Stages (Hand Section) | Baseline (Day 1)
  Assessment will be performed using the hand section of the Brunnström Recovery Stages to classify the stage of motor recovery in the affected hand. The scale has a minimum value of 1 and a maximum value of 6. Higher values indicate better motor function and greater voluntary control of hand movements.
Hand motor control - Brunnström Recovery Stages (Hand Section) | Immediately after therapy completion (Day 15)
  Assessment will be repeated using the Brunnström Recovery Stages to determine any progression in hand motor recovery. The scale has a minimum value of 1 and a maximum value of 6. Higher values indicate better motor function and greater voluntary control of hand movements.